CLINICAL TRIAL: NCT01745146
Title: Anger Self-Management in Post-Acute Traumatic Brain Injury: Clinical Trial
Brief Title: Anger Self-Management in Traumatic Brain Injury
Acronym: ASMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Craig Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tessa Hart, Institute Scientist, MRRI, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 ASMT HN4385; 1R01HD061400-01A2 (NIH)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; TBI; head injury; brain injury; Psych-educational treatment; Anger; irritability; anger management
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anger Self-Management Training (ASMT) (Experimental): 8-session, individual, psycho-educational intervention based on principles of self-monitoring and problem-solving training Significant other (friend or relative) invited to participate in 3 of 8 sessions
  Interventions: Behavioral: ASMT
- Personal Readjustment and Ed (PRE) (Active Comparator): 8-session, individual, psycho-educational intervention based on principles of education and personal readjustment. Significant other (friend or relative) invited to participate in 3 of 8 sessions
  Interventions: Behavioral: PRE

INTERVENTIONS:
Behavioral: ASMT — 8-session, individual, psycho-educational intervention based on principles of self-monitoring and problem-solving training Significant other (friend or relative) invited to participate in 3 of 8 sessions
  Arms: Anger Self-Management Training (ASMT)
Behavioral: PRE — 8-session, individual, psycho-educational intervention based on principles of education and personal readjustment to TBI Significant other (friend or relative) invited to participate in 3 of 8 sessions
  Arms: Personal Readjustment and Ed (PRE)

SUMMARY:
The present study addresses problematic anger and irritability in community dwelling persons with traumatic brain injury (TBI). It is designed to test the worth of a novel treatment approach called Anger Self-Management Training (ASMT), compared to a treatment offering supportive therapy focused on personal readjustment and education, the PRE (Personal Readjustment and Education). The project is a 3-center randomized controlled trial employing equivalent therapist time and therapeutic structure in the delivery of treatment options. The overall aim is to evaluate the relative response rate and correlates of treatment response for the ASMT as compared to the PRE.

DETAILED DESCRIPTION:
Problematic anger/ irritability is common, persistent, and difficult to treat after TBI, and has a broad impact on community and social function. Anger following TBI is related, in part, to deficits in executive function including impaired problem-solving and impaired self-monitoring. In this 2-group, 3-center clinical trial with masked outcome assessment, we will explore feasibility and efficacy of a manualized, 8-session individual treatment, Anger Self-Management Training (ASMT), compared to a treatment using non-specific ingredients of therapist attention, education, and psychological support (PRE).

The ASMT was designed to decrease subjective and objective anger and irritability following traumatic brain injury (TBI), using theoretically motivated "active ingredients." The ASMT focuses on 2 executive deficits implicated in anger post TBI, (1) self-awareness and self-monitoring and (2) problem-solving. Participants will be randomly assigned in 2:1 proportion to ASMT or PRE. The PRE treatment is manualized to the same degree as the ASMT, but focuses on educational and personal readjustment to injury rather than anger-specific strategy training.

The overall goals are to examine the effects of the ASMT compared to PRE on self-reported problematic anger, both 1 week and 2 months after treatment, and to assess the time course of treatment response during the treatment phase.

Specific Aims

1. To examine the efficacy of ASMT compared to a control treatment (PRE) as measured by improvement from baseline to post-treatment on the State-Trait Anger Expression Inventory-Revised (STAXI-2) Trait Anger; STAXI-2 Anger Expression-Out; or the Brief Anger-Aggression Questionnaire (BAAQ) (primary outcome).
2. To examine the trajectory of treatment response within the treatment phase of ASMT/ PRE as shown by a change on 1 or more of the target scales halfway through the treatment (i.e., after 4 of 8 sessions) for those participants who exhibited a positive response post treatment (as defined above).
3. To examine the persistence of treatment effects 2 months after the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 at the time of injury
* ages 18 to 65 at the time of enrollment
* TBI (closed or penetrating) occurring a minimum of 6 months prior to enrollment
* TBI documented as complicated mild, moderate, or severe TBI by any one or more of the following indices:

  * post-resuscitation score on Glasgow Coma Scale (GCS) < 13 or GCS Motor < 6;
  * loss of consciousness, unresponsiveness or coma attributable to the TBI and persisting ≥ 1 hour;
  * post-traumatic amnesia, or disorientation (O x 0, 1 or 2) attributable to the TBI and persisting ≥ 24 hours; or
  * neuro-imaging study positive for TBI-related findings such as contusion, hematoma, hemorrhage, diffuse axonal injury, shear injury, and/ or depressed skull fracture
* Able to travel independently in the community (to maximize the probability that participants will be cognitively and physically able to engage in the treatment)
* Indication from self or other report that participant has problematic anger/ irritability that is new since the injury or worse than before the injury
* Self-report of anger ≥ 1 standard deviation above the mean for age and gender on the Trait Anger or Anger Expression-Out (AX-O) subscales of the State-Trait Anger Expression Inventory-2 (STAXI-2), or a score of ≥ 7 on the Brief Anger-Aggression Questionnaire (BAAQ)
* Able to speak and understand English sufficiently to complete the screening and outcome measures and to participate in a verbally based treatment program, which thus far exists only in English
* Informed consent given by participant or legally authorized representative.

Exclusion Criteria:

* History of schizophrenia or schizo-affective disorder, as documented in medical records or by self-report that a medical professional has given the diagnosis
* Current psychosis, major depression, or suicidal ideation; or history of manic or hypomanic episode as determined by the Mini-International Neuropsychiatric Interview for DSM-IV (MINI) Current alcohol-l dependence, as determined by the MINI.
* Self-reported use of cocaine or amphetamines "daily" or "almost daily" using the relevant questions from the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST)
* TBI requiring hospitalization that has occurred within 6 months prior to enrollment
* Involvement in one-to-one counseling or psychotherapy targeted to emotional health issues
* Involvement in another treatment trial that may affect participation or outcomes
* Evidence of severe, intractable anger as indicated by history of violence-related crimes, e.g., charges for assault.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Hart, PhD, Principal Investigator — Moss Rehabilitation Research Institute
Locations (3):
- United States (3):
  - Craig Hospital, Englewood, Colorado
  - Data Cordinating Center, Englewood, Colorado
  - Moss Rehabilitation Research Institue, Elkins Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hart T, Vaccaro MJ, Hays C, Maiuro RD. Anger self-management training for people with traumatic brain injury: a preliminary investigation. J Head Trauma Rehabil. 2012 Mar-Apr;27(2):113-22. doi: 10.1097/HTR.0b013e31820e686c. PMID 21407088
- [Result] Hart T, Brockway JA, Maiuro RD, Vaccaro M, Fann JR, Mellick D, Harrison-Felix C, Barber J, Temkin N. Anger Self-Management Training for Chronic Moderate to Severe Traumatic Brain Injury: Results of a Randomized Controlled Trial. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):319-331. doi: 10.1097/HTR.0000000000000316. PMID 28520666

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After consent and T1 assessment, participants were randomized (2:1 Anger Self-Management Training or Personal Readjustment and Education) using a computer-generated table provided by the study's Data Coordinating Center, and assigned to the therapist corresponding to their treatment condition. Participants stratified by site.
Groups:
- Personal Readjustment and Education (PRE): Participants provided with education about the effects of traumatic brain injury (TBI) on personal characteristics, relationships, and community roles.
- Anger Self-Management Training (ASMT): Participants provided with education emphasizing the teaching of behavioral skills (self-monitoring, problem-solving) in addition to focused education about anger and its links to traumatic brain injury (TBI).
Period: Overall Study
Arm/Group | Personal Readjustment and Education (PRE) | Anger Self-Management Training (ASMT)
Started | 30 | 60
Allocation to Intervention | 30 | 60
Primary Outcome Assessment | 27 | 57
Analysis | 27 | 57
Completed | 27 | 57
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personal Readjustment and Education (PRE) | Anger Self-Management Training (ASMT) | Total
Number analyzed (Participants) | 30 | 60 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (13.3) | 30.4 (10.2) | 32.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 24 | 49 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 13 | 21
  White | 22 | 40 | 62
  Hispanic or Other | 0 | 7 | 7
Education [Mean (Standard Deviation); unit: years] — Last year of school completed
  years | 13.4 (2.5) | 13.4 (2.1) | 13.4 (2.2)
Cause of Injury [Count of Participants; unit: Participants] — How Traumatic Brain Injury Occurred
  Participants
    Vehicular Incident | 17 | 38 | 55
    Fall | 6 | 8 | 14
    Intentional Injury | 5 | 7 | 12
    Other | 2 | 7 | 9
Median PTA Duration [Count of Participants; unit: Participants] — Median number of days spent in post-traumatic amnesia following TBI. This was ascertained using a structured interview that has been used in other studies of chronic TBI, with the retrospective estimate found to correlate reasonably well with PTA measured prospectively.
  Participants
    < 15 days | 7 | 15 | 22
    15 - 30 days | 9 | 18 | 27
    31 - 90 days | 11 | 15 | 26
    > 90 days | 3 | 12 | 15
Neuropsychological Status [Mean (Standard Deviation); unit: units on a scale] — Intelligence Quotient (IQ) from Wechsler Abbreviated Scale of Intelligence (WASI)Vocabulary and Matrix Reasoning subtests; Range 55-157 (157=best) Rey Auditory Verbal Learning Test (RAVLT) Total; Range 0-75 (75=best) Trail Making Test Part B T-score; Range 7-88 (88=best) Brixton Spatial Anticipation Test error score; Range 0-55 (0=best) Glasgow Outcome Scale-Extended (GOS-E); Range 1-8 (8=best) Global Severity Index (GSI) from the Brief Symptom Inventory (BSI); Range 30-81 (30=best) Frontal Systems Behavior Scale (FrSBe) T-score; Range 9-176 (9=best)
  units on a scale
    IQ Determined from WASI | 94 (16.3) | 97 (16.1) | 95.97 (16.13)
    RAVLT: Sum 5 Trials | 37.8 (9.5) | 40.3 (11.5) | 39.43 (10.9)
    Brixton Spatial Anticipation Test: Error Score | 19.3 (6.7) | 17.2 (7.7) | 17.91 (7.39)
    Trail Making Test Part B: T-Score | 40 (15.2) | 41.2 (13) | 40.81 (13.71)
    GOS-E | 5.6 (0.9) | 6 (1) | 5.87 (0.96)
    BSI GSI | 66.7 (10.3) | 68.9 (8.0) | 68.2 (8.84)
    FrSBe Self-Report | 64.4 (17.4) | 62.4 (15.7) | 63.08 (16.2)
Median Time Post Injury [Median (Full Range); unit: Months] — Number of months between date of injury and start of participation
  Months | 72 [6 to 339] | 69 [6 to 298] | 71 [6 to 339]

OUTCOME MEASURES:

1. Primary Outcome: Post-Treatment Response Rate From Baseline on Anger Measures - Participant Report
Description: Participant report only. The State-Trait Anger Expression Inventory-Revised Trait Anger Scale (STAXI-2 TA) measures how often angry feelings are experienced and the Anger Expression-Out (STAXI-2 AX-O) Scale addresses the expression of anger toward other persons or objects in the environment. The Brief Anger-Aggression Questionnaire (BAAQ) is a 6-item self-report scale that measures frequency of "acting-out" symptoms of anger. Overall treatment response is defined as ≥ 1 standard deviation change in the direction of improvement from pre- to 10 wk post-treatment on any 1 of the three anger scales used. Analysis first done by including participants who did not complete the assessment as non-responders (labeled as "missing outcomes included" or "MOI"). Analysis done a second time only using participants who completed the assessment (labeled as "missing outcomes removed" or "MOR").
Time Frame: Baseline, 10 weeks (post-treatment)
Population: Missing outcomes originally treated as non-Responders (Protocol Specified) and then taken out of data set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Difference: The difference in treatment response rates between the ASMT group and the PRE group.
Arm/Group | Personal Readjustment and Education (PRE) | Anger Self-Management Training (ASMT) | Difference
Number analyzed (Participants) | 30 | 60 | 90
percentage of participants
  STAXI-2 TA (MOI) | 46.7 [28.9 to 64.6] | 68.3 [56.5 to 80.1] | 21.7 [0.3 to 41.8]
  STAXI-2 AX-O (MOI) | 50.0 [32.1 to 68.0] | 56.7 [44.2 to 69.2] | 6.7 [-14.6 to 27.7]
  BAAQ (MOI) | 16.7 [3.4 to 30.0] | 11.7 [3.2 to 19.1] | -5.0 [-22.2 to 8.4]
  Overall (MOI) | 63.3 [46.0 to 80.1] | 71.1 [60.3 to 83.1] | 8.3 [-11.1 to 29.0]
  STAXI-2 TA (MOR): number analyzed (Participants) | 27 | 57 | 84
  STAXI-2 TA (MOR) | 51.9 [33.0 to 70.8] | 71.9 [60.2 to 83.6] | 20.1 [-1.6 to 41.2]
  STAXI-2 AX-O (MOR): number analyzed (Participants) | 27 | 57 | 84
  STAXI-2 AX-O (MOR) | 55.6 [36.9 to 74.3] | 59.6 [46.9 to 72.3] | 4.1 [-17.5 to 26.3]
  BAAQ (MOR): number analyzed (Participants) | 27 | 57 | 84
  BAAQ (MOR) | 18.5 [3.8 to 33.1] | 12.3 [3.8 to 20.8] | -6.2 [-24.8 to 8.2]
  Overall (MOR): number analyzed (Participants) | 27 | 57 | 84
  Overall (MOR) | 70.4 [53.2 to 87.6] | 75.4 [64.2 to 86.6] | 5.1 [-13.5 to 26.3]
Statistical Analysis 1: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for STAXI-2 Trait Anger. Missing outcomes reported at non-responders; Test type: Equivalence — Primary outcome is difference in rates of treatment response between the ASMT and the PRE, where treatment response is defined as ≥ 1 SD improvement in self-reported anger on at least 1 of 3 target scales from pre- to 1-2 wk post treatment. The treatment will be considered supported if the observed response rate with ASMT is at least 20 percentage points higher than that with the control treatment, PRE; p = 0.047, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 2: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for STAXI-2 Anger Expression-Out. Missing outcomes reported at non-responders; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.549, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 3: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for BAAQ. Missing outcomes reported at non-responders; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.511, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 4: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for STAXI-2 Trait Anger. Missing outcomes excluded for this analysis; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.031, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 5: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for STAXI-2 Anger Expression-Out. Missing outcomes excluded for this analysis; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.483, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 6: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in post-treatment response rate for BAAQ. Missing outcomes excluded for this analysis; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.530, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's chi-square test
Statistical Analysis 7: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in overall post-treatment response rate. Missing outcomes included as non-responders; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.421, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's Chi-squared
Statistical Analysis 8: Comparison: Personal Readjustment and Education (PRE) vs Anger Self-Management Training (ASMT); Significance of difference in overall post-treatment response rate. Missing outcomes excluded for this analysis; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.332, Chi-squared — Alpha was set at .05 both for the a priori hypotheses and also for secondary analyses; Pearson's Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored from the first treatment session to the final outcome evaluation. This consisted of a monitoring period of 4 months per study participant. Adverse events (AE) and serious adverse events (SAE) were queried with a checklist at each data collection episode and each therapy session through study completion (4 months altogether). If endorsed, events were evaluated as to seriousness, duration, resolution date if any, and possible relationship to study procedures.
Description: For SAEs, we adhered to a standard definition used in medical trials: any event for which the outcome is death, hospitalization, life-threatening (i.e., person is at risk of death at the time of the event) or the event leads to disability and/or incapacity, or requires intervention to prevent those outcomes. We defined AEs as self-reported emergency care visits, arrests, episodes of violence, thoughts of harming self or others and withdrawal from therapy sessions and/or from the study at large.
Arm/Group | Personal Readjustment and Education (PRE) | Anger Self-Management Training (ASMT)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/30 | 7/60
Other Adverse Events (participants affected / at risk) | 9/30 | 2/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personal Readjustment and Education (PRE) (N=30) | Anger Self-Management Training (ASMT) (N=60)
Admission to Hospital or Overnight Treatment Facility (Surgical and medical procedures) | 2 (2) | 7 (7) — Involved admission to a hospital or other overnight treatment facility, most often for planned procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personal Readjustment and Education (PRE) (N=30) | Anger Self-Management Training (ASMT) (N=60)
Episode of rage (Psychiatric disorders) | 9 (9) | 2 (2)

LIMITATIONS AND CAVEATS:
All participants had self-reported problems with anger and were excluded for serious limitations in communication. Thus, the study cannot be generalized to those with very severe cognitive or communication deficits or who deny anger problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No